CLINICAL TRIAL: NCT00002582
Title: UKCCCR RANDOMISED TRIAL OF ADJUVANT ENDOCRINE THERAPY AND CHEMOTHERAPY IN WOMEN WITH EARLY BREAST CANCER, THE ADJUVANT BREAST CANCER (ABC) TRIAL
Brief Title: Tamoxifen, Ovarian Ablation, and/or Chemotherapy in Treating Women With Stage I, Stage II, or Stage IIIA Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research Campaign Clinical Trials Centre (Other); Scottish Cancer Therapy Network (Other); Yorkshire Regional Clinical Trials Research Unit (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NCRI-ABC; CDR0000063697 (Registry Identifier: PDQ (Physician Data Query)); CRC-TU-BR3010; SCTN-BR9401/BR9402; YRCO-ABC; EU-94029; UKCCCR-ABC
Record Dates: First submitted 1999-11-01; First posted 2003-07-08 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CMF regimen; Cyclophosphamide; Doxorubicin; Fluorouracil; Goserelin; Leuprolide; Methotrexate; Tamoxifen; Ovariectomy; Radiotherapy

INTERVENTIONS:
Drug: CMF regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: fluorouracil
Drug: goserelin acetate
Drug: leuprolide acetate
Drug: methotrexate
Drug: tamoxifen citrate
Procedure: oophorectomy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen. Combination chemotherapy uses different ways to stop tumor cells from dividing so they stop growing or die. Combining hormone therapy with chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of tamoxifen with or without chemotherapy and/or ovarian ablation in treating women with stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate overall and relapse-free survival of women with early-stage breast cancer receiving adjuvant tamoxifen with or without adjuvant chemotherapy and/or ovarian suppression.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by participating institution and choice of randomization option.

Postmenopausal women are randomized to the first or second groups.

Randomization for pre- and perimenopausal women is based on the clinician's judgement of appropriate adjuvant therapy (chemotherapy and/or ovarian suppression). Patients may be randomized as follows: among all four groups; for chemotherapy alone (first versus second group); for ovarian suppression alone (first versus third group); for ovarian suppression with nonrandomized assignment to chemotherapy (second versus forth group); for chemotherapy with nonrandomized assignment to ovarian suppression (second versus fourth group).

* First group: Patients receive tamoxifen by mouth every day for 5 years.
* Second group: Patients receive tamoxifen plus cyclophosphamide, methotrexate, fluorouracil (CMF) or doxorubicin/cyclophosphamide (AC). CMF is given every month for 6 courses; AC is given every 3 weeks for 4 courses.
* Third group: Patients receive tamoxifen plus ovarian suppression by oophorectomy, radiation castration, or leuprolide or goserelin.
* Fourth group: Patients receive tamoxifen plus ovarian suppression plus chemotherapy with CMF or AC.

Patients are followed for overall and relapse-free survival.

PROJECTED ACCRUAL: Approximately 6,000 women (4,000 premenopausal, 2,000 postmenopausal) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive carcinoma of the breast for which adjuvant systemic therapy is appropriate

  * Stage I, II, or IIIA
  * Pathologically positive or negative nodes
  * Any size primary tumor
* No edema, peau d'orange, infiltration of the skin, or direct extension to the chest wall
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Pre-, peri-, or postmenopausal

Performance status:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior malignancy except:

  * Basal cell carcinoma
  * Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior systemic treatment for breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 1993-06; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Yarnold, MD, FRCR, Study Chair — Royal Marsden NHS Foundation Trust; Helena Earl, MBBS, PhD, FRCP, Study Chair — Cancer Research Campaign Clinical Trials Centre; Stanley B. Kaye, MD, FRCP, Study Chair — University of Glasgow; Tim J. Perren, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (2):
- United Kingdom (2):
  - Cancer Research Campaign Trials Unit-Birmingham (CRCTU), Birmingham, England
  - Beatson Oncology Centre, Glasgow, Scotland

REFERENCES:
- [Background] Perren TJ. Adjuvant therapy for operable breast cancer; more answers, new questions. Br J Cancer. 1995 Jun;71(6):1142-4. doi: 10.1038/bjc.1995.223. No abstract available. PMID 7779702
- [Background] Brunt AM. The UKCCCR adjuvant breast cancer (ABC) trial. ABC Trial Steering Committee. Clin Oncol (R Coll Radiol). 1994;6(4):209-10. doi: 10.1016/s0936-6555(05)80287-0. No abstract available. PMID 7986756
- [Background] Yarnold JR, Bliss JM, Brunt M, Earl H, Kaye S, Mason M, Mossman J, Perren T, Richards M. Management of breast cancer. Refer women to multidisciplinary breast clinics. BMJ. 1994 Mar 12;308(6930):714-5. doi: 10.1136/bmj.308.6930.714a. No abstract available. PMID 8142803
- [Background] Bliss JM, Yarnold JR. Treatment of early breast cancer. Lancet. 1992 Apr 11;339(8798):936. doi: 10.1016/0140-6736(92)90981-8. No abstract available. PMID 1348335
- [Result] Adjuvant Breast Cancer Trials Collaborative Group. Polychemotherapy for early breast cancer: results from the international adjuvant breast cancer chemotherapy randomized trial. J Natl Cancer Inst. 2007 Apr 4;99(7):506-15. doi: 10.1093/jnci/djk108. PMID 17405995
- [Result] Adjuvant Breast Cancer Trials Collaborative Group. Ovarian ablation or suppression in premenopausal early breast cancer: results from the international adjuvant breast cancer ovarian ablation or suppression randomized trial. J Natl Cancer Inst. 2007 Apr 4;99(7):516-25. doi: 10.1093/jnci/djk109. PMID 17405996